CLINICAL TRIAL: NCT02538484
Title: A Phase 0, Investigator Initiated Study, Evaluating the Impact of Omega 3 Fatty Acid Supplementation on Aromatase in Obese Postmenopausal Women With Estrogen Receptor Positive Breast Cancer
Brief Title: Impact of Omega 3 Fatty Acid Supplementation on Aromatase in Obese Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTMS# 15-2100; HSC20150602H (Other: UT Health Science Center Institutional Review Board)
Record Dates: First submitted 2015-08-11; First posted 2015-09-02 (Estimated); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Letrozole (Active Comparator): Letrozole 2.5 mg by mouth daily for 30 days.
  Interventions: Drug: Letrozole
- Fish Oil (Active Comparator): Fish oil 2700 mg by mouth daily for 30 days.
  Interventions: Dietary Supplement: Fish Oil
- Letrozole and Fish Oil (Active Comparator): Letrozole 2.5 mg and Fish oil 2700 mg by mouth daily for 30 days.
  Interventions: Drug: Letrozole; Dietary Supplement: Fish Oil

INTERVENTIONS:
Drug: Letrozole — Aromatase inhibitor
  Other Names: Femara
  Arms: Letrozole; Letrozole and Fish Oil
Dietary Supplement: Fish Oil — Omega-3 free fatty acid
  Other Names: Omega-3
  Arms: Fish Oil; Letrozole and Fish Oil

SUMMARY:
Assess the impact of dietary omega 3 free fatty acids and/or letrozole on obese, postmenopausal breast cancer patients.

DETAILED DESCRIPTION:
Prospective, comparative, three arm, short term, non-interventional study with correlative biomarker endpoints. Sixty (60) obese (≥ 30 BMI) newly diagnosed ER+ postmenopausal breast cancer patients will be recruited to participate in a short term (30 day) Phase 0 biomarker evaluation study prior to surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Postmenopausal as confirmed in medical history
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB (Institutional Review Board)/Ethics Committee.
* Estrogen receptor positive breast cancer. Body mass index of 30 or greater.
* Consented for tissue collection on CTRC (Cancer Therapy and Research Center) repository 07-32

Exclusion Criteria:

* Cachexia
* Active systemic illness (infection including viral illnesses such as Hepatitis and HIV)
* Chronic use of NSAIDs (nonsteroidal anti-inflammatory drugs) aspirin or omega-3 free fatty acid supplementation within the last 60 days (defined as greater than or equal to 7 consecutive days)
* Any NSAIDs aspirin or omega-3 free fatty acid supplementation within the last 14 days
* History of medical noncompliance
* Scheduled date of surgical resection that would limit the amount of time taking the intervention to less than 21 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Change in levels of aromatase target gene. | 30 Days
Change in serum levels of PGE2 (prostaglandin E2). | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, MD, PhD, Principal Investigator — Principal Investigator
Locations (2):
- United States (2):
  - Houston Methodist Cancer Center at Texas Medical Center, Houston, Texas
  - Mays Cancer Center, UT Health San Antonio, San Antonio, Texas